CLINICAL TRIAL: NCT01656252
Title: Phase I Dose Finding/Phase II Placebo-Controlled Trial of Eltrombopag During Consolidation Therapy in Adults With Acute Myeloid Leukemia (AML) in Complete Remission
Brief Title: Trial of Eltrombopag During Consolidation Therapy in Adults With AML in Complete Remission
Acronym: PrE0901
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study stopped per Novartis request due to futility from another study.
Sponsor: PrECOG, LLC. (Other)
Collaborators: GlaxoSmithKline (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PrE0901; ELT114465 (Other Grant/Funding Number: GSK/Novartis)
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Leukemia; Complete Remission; Consolidation; Consolidation Chemotherapy; Cytarabine; Eltrombopag; Leukemia; Thrombocytopenia; Thrombopoietin
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Pathologic Complete Response; Leukemia; Thrombocytopenia; Jacobs syndrome | interventions — eltrombopag; Cytarabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase I- Cytarabine & Eltrombopag (Experimental): Cycle 1= Cytarabine twice daily on Days 1, 3 and 5 and Eltrombopag (Open-Label) until platelet recovery or for 35 consecutive days, whichever occurs first. Phase I will determine the dose and schedule of Eltrombopag to be used in Phase II.
  Interventions: Drug: Phase I- Cytarabine & Eltrombopag
- Phase II- Sequence A (Experimental): Cytarabine twice daily on Days 1, 3 and 5. Eltrombopag(dose and schedule as determined in Phase I) with 1st cycle of high-dose consolidation chemotherapy and placebo with 2nd cycle. Treatment sequence will be blinded to the patient and all study/sponsor personnel.
  Interventions: Drug: Phase II- Sequence A
- Phase II- Sequence B (Experimental): Cytarabine twice daily on Days 1, 3 and 5. Placebo with 1st cycle of high-dose consolidation therapy and Eltrombopag(dose and schedule as determined in Phase I) with 2nd cycle. Treatment sequence will be blinded to the patient and all study/sponsor personnel.
  Interventions: Drug: Phase II- Sequence B

INTERVENTIONS:
Drug: Phase I- Cytarabine & Eltrombopag — Cycle 1= Cytarabine 3 g/m² IV twice daily on Days 1, 3 and 5 (Patients >60 years of age will receive cytarabine 1.5 g/m² IV per dose). Day 1 must start in AM.
  Eltrombopag (Open-Label) by mouth daily until platelet recovery or for 35 consecutive days, whichever occurs first. Phase I will determine the dose and schedule of Eltrombopag to be used in Phase II.
  One cycle of consolidation therapy with high-dose cytarabine and eltrombopag will be received on study. Additional chemotherapy may be administered at the investigators discretion without eltrombopag.
  Other Names: Ara-C; Cytosar-U; Cytosine Arabinoside; Promacta; Thrombopoietic Agent
  Arms: Phase I- Cytarabine & Eltrombopag
Drug: Phase II- Sequence A — Cytarabine 3 g/m² IV twice daily on Days 1, 3 and 5 (Patients >60 years of age will receive cytarabine 1.5 g/m² IV per dose). Day 1 must start in AM.
  Eltrombopag by mouth daily (dose and schedule as determined in Phase I) with 1st cycle of high-dose consolidation chemotherapy and placebo by mouth daily with 2nd cycle.
  Eltrombopag/placebo will continue until platelet recovery or for 35 consecutive days, whichever occurs first.
  Additional chemotherapy may be administered at the investigators discretion without eltrombopag.
  Other Names: Ara-C; Cytosar-U; Cytosine Arabinoside; Promacta; Thrombopoietic Agent
  Arms: Phase II- Sequence A
Drug: Phase II- Sequence B — Cytarabine 3 g/m² IV twice daily on Days 1, 3 and 5 (Patients >60 years of age will receive cytarabine 1.5 g/m² IV per dose). Day 1 must start in AM.
  Placebo by mouth daily with 1st cycle of high-dose consolidation therapy and Eltrombopag by mouth daily (dose and schedule as determined in Phase I) with 2nd cycle.
  Eltrombopag/placebo will continue until platelet recovery or for 35 consecutive days, whichever occurs first.
  Additional chemotherapy may be administered at the investigators discretion without eltrombopag.
  Other Names: Ara-C; Cytosar-U; Cytosine Arabinoside; Promacta; Thrombopoietic Agent
  Arms: Phase II- Sequence B

SUMMARY:
Patients with Acute Myeloid Leukemia (AML) in complete remission will receive eltrombopag while undergoing consolidation chemotherapy with high-dose cytarabine. Eltrombopag may help increase the number of platelets during chemotherapy and may help prevent the risk of bleeding.

Phase I will study the side effects, best dose and platelet effects of eltrombopag when given with consolidation chemotherapy. After the maximum safe and tolerated dose and schedule is found in Phase I, the study will proceed to Phase II. Phase II will confirm the dose and schedule of eltrombopag identified in Phase I that can increase platelet counts in patients receiving consolidation therapy.

DETAILED DESCRIPTION:
Consolidation chemotherapy with high dose cytarabine usually causes myelosuppression for 14 to 21 days after each treatment. Patients have low blood counts for days or weeks before the bone marrow resumes function. This may result in e.g., hospitalization, treatment with antibiotics, and transfusions with blood and/or platelets. In addition, this may cause a delay in treatment and reduction in dose. To achieve the best outcome from treatment, dose reductions and delays in treatment must be avoided.

The incidence and duration of decreased white blood cells (neutropenia) and neutropenic complications have been reduced by the use of growth colony stimulating factors. Additionally, the use of erythropoietin-stimulating factors has reduced anemia and the need for red blood cell transfusions. Thrombocytopenia remains an important limiting factor in administration of chemotherapy and maintaining dose intensity in some patients. Additionally, the risk of bleeding secondary to low platelet counts may increase sickness or even death in patients undergoing cancer treatment.

Thrombopoietin (TPO) is the principal cytokine involved in the regulation of megakaryopoiesis and platelet production. Eltrombopag is an orally bioavailable, small molecule, TPO-receptor agonist that stimulates platelet production by a similar, but not identical, mechanism to endogenous TPO. Eltrombopag has been approved in the U.S. for the treatment of chronic Idiopathic Thrombocytopenic Purpura. Eltrombopag is also under development for other indications such as Hepatitis C Virus-associated thrombocytopenia, Myelodysplastic Syndrome/AML, and oncology related thrombocytopenias. This agent appears to possess many of the desirable properties for a treatment for chemotherapy induced thrombocytopenia, including oral administration.

The Phase I portion of this study will be conducted using a dose escalation/de-escalation strategy for patients in either the first or second complete remission. Dose escalations are planned in the form of both acceleration of date of initiation of eltrombopag relative to the start of consolidation chemotherapy as well as increasing daily dosing.

The Phase II portion will be conducted using the dose and schedule selected from the Phase I portion of the study for those patients in first complete remission. Patients will be used as their own controls, e.g., a two-period two-treatment cross-over design. Patients will be randomly allocated 1:1 to one of two sequences. Patients randomized to Sequence A will receive eltrombopag with their first cycle of consolidation and placebo with Cycle 2. Patients randomized to Sequence B will receive placebo with their first cycle of consolidation and eltrombopag with Cycle 2. The treatment assignment will be blinded to the patient and all study/sponsor personnel.

Patients will undergo blood sample collection for Thrombopoietin(TPO)/ Erythropoietin(EPO) and pharmacokinetic analysis of eltrombopag in Phase I and pharmacokinetic analysis of eltrombopag in the Phase II portion of the study.

ELIGIBILITY:
Inclusion Criteria:

• Cytomorphologically documented diagnosis of acute myeloid leukemia (AML). Acute promyelocytic leukemia patients will be excluded (FAB M3). FAB classification, cytogenetics and molecular markers (if applicable) must be available at registration.

Phase I Enrollment:

* Must be in first or second complete remission, e.g., no evidence of active disease in blood, bone marrow (<5% blasts), or other tissues.
* For each remission, may have received no more than 2 cycles of induction treatment (any type).
* May have received no more than one course of consolidation for the current remission prior to enrollment (any type)

Phase II Enrollment:

* Must be in first complete remission, e.g., no evidence of active disease in blood, bone marrow (<5% blasts), or other tissues.
* May have received no more than 2 cycles of induction treatment (any type).

Enrollment in Either Phase:

* Remission status must be documented by a bone marrow examination up to 28 days prior to study registration.
* Have recovered from induction and first consolidation (if applicable) therapy side effects (or ≤grade 1).
* ≥18 years of age and ≤70 years of age.
* ECOG performance status 0, 1, 2.
* Have not received cytotoxic drug therapy within 21 days of registration.
* Have not received hematopoietic colony stimulating growth factors within 14 days of registration.
* Have not received packed red blood cells or platelets within 7 days of registration.
* Have not received investigational agents within 30 days of registration and will not receive any investigational agents other than eltrombopag/placebo during study.
* Signed IRB-approved informed consent.
* Willing to provide blood samples for research purposes.
* Adequate organ function obtained within 28 days prior to registration:

  * Absolute neutrophil count >1 x 10⁹/L
  * Platelet count >100 x 10⁹/L
  * Total direct serum bilirubin ≤1.5x upper limit of normal (ULN)
  * ALT and AST ≤3x ULN
  * BUN and serum creatinine <2x ULN
  * Albumin ≥2.5 g/dL
  * PT and PTT 80-120% of institutional normal range
* Women of childbearing potential must have a negative serum pregnancy test within 14 days of registration.
* Not pregnant nor breast feeding.
* Women of childbearing potential and sexually active males must use an accepted and effective method of contraception.
* Patients of known East Asian ancestry (Chinese, Japanese, Taiwanese, and Korean) are excluded from protocol participation for safety and efficacy reasons.
* Able to swallow and retain orally administered medication.
* No clinically significant gastrointestinal abnormalities such as malabsorption syndrome or major resection of the stomach or bowels.
* No clinical evidence of hepatomegaly or splenomegaly.
* No known risk for Torsades de Pointes. (Eltrombopag use has not been shown to be associated with Torsades de Pointes.)
* No active or unresolved infection and must be off all antibiotics for at least 7 days prior to registration.
* No current evidence of invasive fungal infection.
* No known Hepatitis B, Hepatitis C active disease.
* No known Human Immunodeficiency Virus (HIV) seropositivity. The risk for potential toxicities secondary to HIV (e.g., increased risk for fatal opportunistic infection) may confound the toxicity profile of eltrombopag.
* Patients with a history of Central Nervous System (CNS) leukemia are eligible if there is documentation of no current CNS involvement on cerebrospinal fluid (CSF) examination (e.g., negative CSF by lumbar puncture) within 28 days of registration.
* No prior or concomitant malignancy in the past 5 years which is currently active and likely to interfere with the patient's treatment for AML or which is likely to increase the patient's morbidity or mortality. No prior chemotherapy or radiation therapy allowed (unless related to AML treatment).
* No concurrent organ damage or medical problems that would prohibit therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hillard M Lazarus, MD, Study Chair — University Hospitals Cleveland Medical Center
Locations (5):
- United States (5):
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Data is proprietary.

REFERENCES:
- [Background] Mavroudi I, Pyrovolaki K, Pavlaki K, Kozana A, Psyllaki M, Kalpadakis C, Pontikoglou C, Papadaki HA. Effect of the nonpeptide thrombopoietin receptor agonist eltrombopag on megakaryopoiesis of patients with lower risk myelodysplastic syndrome. Leuk Res. 2011 Mar;35(3):323-8. doi: 10.1016/j.leukres.2010.06.029. Epub 2010 Aug 4. PMID 20688394
- [Background] Will B, Kawahara M, Luciano JP, Bruns I, Parekh S, Erickson-Miller CL, Aivado MA, Verma A, Steidl U. Effect of the nonpeptide thrombopoietin receptor agonist Eltrombopag on bone marrow cells from patients with acute myeloid leukemia and myelodysplastic syndrome. Blood. 2009 Oct 29;114(18):3899-908. doi: 10.1182/blood-2009-04-219493. Epub 2009 Aug 26. PMID 19710504
- [Background] Kellum A, Jagiello-Gruszfeld A, Bondarenko IN, Patwardhan R, Messam C, Mostafa Kamel Y. A randomized, double-blind, placebo-controlled, dose ranging study to assess the efficacy and safety of eltrombopag in patients receiving carboplatin/paclitaxel for advanced solid tumors. Curr Med Res Opin. 2010 Oct;26(10):2339-46. doi: 10.1185/03007995.2010.510051. PMID 20735290
- [Background] Vadhan-Raj S. Management of chemotherapy-induced thrombocytopenia: current status of thrombopoietic agents. Semin Hematol. 2009 Jan;46(1 Suppl 2):S26-32. doi: 10.1053/j.seminhematol.2008.12.007. PMID 19245931
- [Result] Strickland SA, Wang XV, Cerny J, Rowe JM, Rybka W, Tallman MS, Litzow M, Lazarus HM. A novel PrECOG (PrE0901) dose-escalation trial using eltrombopag: enhanced platelet recovery during consolidation therapy in acute myeloid leukemia. Leuk Lymphoma. 2020 Sep;61(9):2191-2199. doi: 10.1080/10428194.2020.1762878. Epub 2020 May 30. PMID 32476546

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study closed after phase I. Phase II study was not conducted.
Pre-assignment Details: One patient did not start treatment because of an infection before starting protocol treatment.
Groups:
- Phase I- Cytarabine & Eltrombopag: Cycle 1= Cytarabine twice daily on Days 1, 3 and 5 and Eltrombopag (Open-Label) until platelet recovery or for 35 consecutive days, whichever occurs first. Phase I will determine the dose and schedule of Eltrombopag to be used in Phase II.
  Phase I- Cytarabine & Eltrombopag: Cycle 1= Cytarabine 3 g/m² IV twice daily on Days 1, 3 and 5 (Patients >60 years of age will receive cytarabine 1.5 g/m² IV per dose). Day 1 must start in AM.
  Eltrombopag (Open-Label) by mouth daily until platelet recovery or for 35 consecutive days, whichever occurs first. Phase I will determine the dose and schedule of Eltrombopag to be used in Phase II.
  One cycle of consolidation therapy with high-dose cytarabine and eltrombopag will be received on study. Additional chemotherapy may be administered at the investigators discretion without eltrombopag.
Period: Phase I
Arm/Group | Phase I- Cytarabine & Eltrombopag
Started | 14
Completed | 14
Not Completed | 0
Period: Phase II
Arm/Group | Phase I- Cytarabine & Eltrombopag
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligible, treated patients
Arm/Group | Phase I- Cytarabine & Eltrombopag
Number analyzed (Participants) | 14
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [49 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Phase I- Optimal Tolerated Dose of Eltrombopag
Description: To determine the safety, tolerability and optimal dose of eltrombopag in acute myeloid leukemia patients in complete remission receiving intensive consolidation chemotherapy. The optimal dose was based on rules involving observation of Dose Limiting Toxicity (DLT events), defined as a CTCAE Version 4 non-hematologic adverse event of grade 3 or higher occurring within 30 days of the last dose of eltrombopag judged by the investigator to be at least possibly related to eltrombopag administration.
Time Frame: 13 months
Measure: Number; unit: mg
Arm/Group | Phase I- Cytarabine & Eltrombopag
Number analyzed (Participants) | 14
mg | 300

2. Primary Outcome: Phase I - Dose Level With Best Kinetics of Platelet Count Recovery
Description: To describe the kinetics of platelet count recovery in acute myeloid leukemia patients in complete remission receiving intensive consolidation chemotherapy who will be receiving eltrombopag. This is assessed graphically by plotting platelet count vs. days relative to start of cytarabine for each patient.
Time Frame: 13 months
Measure: Number; unit: mg
Arm/Group | Phase I- Cytarabine & Eltrombopag
Number analyzed (Participants) | 14
mg | 150

3. Primary Outcome: Phase II- Assess if Platelet Count Recovery is Increased With Eltrombopag
Description: To determine if platelet recovery following consolidation chemotherapy is accelerated with eltrombopag.
Time Frame: 62 months
Population: Study terminated during Phase I. No Phase II patients enrolled.
Groups:
- Phase II- Sequence A: Cytarabine twice daily on Days 1, 3 and 5. Eltrombopag(dose and schedule as determined in Phase I) with 1st cycle of high-dose consolidation chemotherapy and placebo with 2nd cycle. Treatment sequence will be blinded to the patient and all study/sponsor personnel.
  Phase II- Sequence A: Cytarabine 3 g/m² IV twice daily on Days 1, 3 and 5 (Patients >60 years of age will receive cytarabine 1.5 g/m² IV per dose). Day 1 must start in AM.
  Eltrombopag by mouth daily (dose and schedule as determined in Phase I) with 1st cycle of high-dose consolidation chemotherapy and placebo by mouth daily with 2nd cycle.
  Eltrombopag/placebo will continue until platelet recovery or for 35 consecutive days, whichever occurs first.
  Additional chemotherapy may be administered at the investigators discretion without eltrombopag.
- Phase II- Sequence B: Cytarabine twice daily on Days 1, 3 and 5. Placebo with 1st cycle of high-dose consolidation therapy and Eltrombopag(dose and schedule as determined in Phase I) with 2nd cycle. Treatment sequence will be blinded to the patient and all study/sponsor personnel.
  Phase II- Sequence B: Cytarabine 3 g/m² IV twice daily on Days 1, 3 and 5 (Patients >60 years of age will receive cytarabine 1.5 g/m² IV per dose). Day 1 must start in AM.
  Placebo by mouth daily with 1st cycle of high-dose consolidation therapy and Eltrombopag by mouth daily (dose and schedule as determined in Phase I) with 2nd cycle.
  Eltrombopag/placebo will continue until platelet recovery or for 35 consecutive days, whichever occurs first.
  Additional chemotherapy may be administered at the investigators discretion without eltrombopag.
Arm/Group | Phase I- Cytarabine & Eltrombopag | Phase II- Sequence A | Phase II- Sequence B
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Phase I & Phase II- Pharmacokinetics of Eltrombopag
Description: To determine the plasma concentrations of eltrombopag in acute myeloid leukemia patients in complete remission receiving intensive consolidation chemotherapy (selected dosing regimen only).
Time Frame: 62 months
Population: Data was not collected.
Arm/Group | Phase I- Cytarabine & Eltrombopag | Phase II- Sequence A | Phase II- Sequence B
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Phase II- Platelet Transfusion Requirements
Description: To determine the impact of eltrombopag on platelet transfusion requirements in the setting of consolidation chemotherapy.
Time Frame: 62 months
Population: Study terminated during Phase I. No Phase II patients enrolled.
Arm/Group | Phase I- Cytarabine & Eltrombopag | Phase II- Sequence A | Phase II- Sequence B
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Phase II- Red Blood Cell Transfusion Requirements
Description: To determine the impact of eltrombopag on red blood cell transfusion requirements.
Time Frame: 62 months
Population: Study terminated during Phase I. No Phase II patients enrolled.
Arm/Group | Phase I- Cytarabine & Eltrombopag | Phase II- Sequence A | Phase II- Sequence B
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Phase II- Bleeding Event Occurrence
Description: To determine the impact of eltrombopag on occurrence of bleeding events.
Time Frame: 62 months
Population: Study terminated during Phase I. No Phase II patients enrolled.
Arm/Group | Phase I- Cytarabine & Eltrombopag | Phase II- Sequence A | Phase II- Sequence B
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Phase II- Time to Platelet Count Recovery
Description: To determine the impact of eltrombopag on time to platelet recovery following consolidation chemotherapy.
Time Frame: 62 months
Population: Study terminated during Phase I. No Phase II patients enrolled.
Arm/Group | Phase I- Cytarabine & Eltrombopag | Phase II- Sequence A | Phase II- Sequence B
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Phase II- Depth of Platelet Nadir
Description: To determine the impact of eltrombopag on the depth of platelet nadir following a cycle of consolidation chemotherapy.
Time Frame: 62 months
Population: Study terminated during Phase I. No Phase II patients enrolled.
Arm/Group | Phase I- Cytarabine & Eltrombopag | Phase II- Sequence A | Phase II- Sequence B
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Phase II- Duration of Platelet Nadir
Description: To determine the duration of platelet nadir in the setting of eltrombopag exposure.
Time Frame: 62 months
Population: Study terminated during Phase I. No Phase II patients enrolled.
Arm/Group | Phase I- Cytarabine & Eltrombopag | Phase II- Sequence A | Phase II- Sequence B
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Phase II- Safety of Eltrombopag With Consolidation
Description: To determine the safety and tolerability of eltrombopag when given at the optimal dose in the setting of consolidation chemotherapy.
Time Frame: 62 months
Population: Study terminated during Phase I. No Phase II patients enrolled.
Arm/Group | Phase I- Cytarabine & Eltrombopag | Phase II- Sequence A | Phase II- Sequence B
Number analyzed (Participants) | 0 | 0 | 0

12. Other Pre Specified Outcome: Exploratory- Eltrombopag Effect on TPO/EPO
Description: To determine if eltrombopag has an effect on TPO and/or EPO in this setting.
Time Frame: 62 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Participants were assessed by the clinician at every treatment cycle while on treatment and for 30 days after the end of treatment.
Arm/Group | Phase I- Cytarabine & Eltrombopag
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 10/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I- Cytarabine & Eltrombopag (N=14)
Anemia (Blood and lymphatic system disorders) | 2
Platelet Count Decreased (Investigations) | 1
Neutrophil Count Decreased (Investigations) | 2
Alanine Aminotransferase Increased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 1
Blood Bilirubin Increased (Investigations) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Investigations) | 2
Dizziness (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 7
Flu Like Symptoms (General disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Menorrhagia (Reproductive system and breast disorders) | 1
Mucositis Oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No